CLINICAL TRIAL: NCT06148259
Title: Comparison of Two Novel Anti Diabetes Medications Classes as Regard Prostate Symptoms in Patient With Diabetes
Brief Title: SGLT Inhibitors Versus DDP4 Inhibitors and Prostate in Patient With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor of Internal medicine and nephrology, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N-136-2023
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Prostatic Hyperplasia
MeSH Terms: conditions — Diabetes Mellitus; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium glucose cotransporter 2 inhibitors (Active Comparator): patients with diabetes treated with sodium glucose cotransporter 2- Dapagliflozin
  Interventions: Other: International prostate symptom score; Diagnostic Test: Assessment of prostate volume; Other: Pittsburgh sleep quality Index; Diagnostic Test: Glycated hemoglobin
- Dipeptidyl peptidase 4 inhibitors (Active Comparator): patients with diabetes treated with Dipeptidyl peptidase 4 inhibitor-sitagliptin
  Interventions: Other: International prostate symptom score; Diagnostic Test: Assessment of prostate volume; Other: Pittsburgh sleep quality Index; Diagnostic Test: Glycated hemoglobin

INTERVENTIONS:
Other: International prostate symptom score — Questionnaire of 8 questions to be administered to all patients about prostate symptoms
Diagnostic Test: Assessment of prostate volume — Measurements using ultrasound
Other: Pittsburgh sleep quality Index — Questionnaire to assess quality of sleep
Diagnostic Test: Glycated hemoglobin — Measures control of diabetes

SUMMARY:
The study aims to compare the effect of two different classes of anti- diabetes medications on prostate volume and symptoms in elderly patients with diabetes mellitus

DETAILED DESCRIPTION:
The study aims to compare the effect of two different classes of anti- diabetes medications on prostate volume and symptoms in elderly patients with diabetes mellitus The study compares sodium glucose cotransporter 2 inhibitors to Dipeptidyl peptidase 4 inhibitors in elderly patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes and benign prostatic hyperplasia should be on monotherapy with either SGLT inhibitor or DDP4 inhibitors

Exclusion Criteria:

* unable to consent to the blood sampling or ultrasound Any other diabetes control measure other than SGLT inhibitors or DDP 4 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with benign prostatic hyperplasia
Enrollment: 57 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
change in prostate volume | one year
  The delta change in prostate volume as measured by Ultrasound
Change in prostate symptoms | one year
  As indicated by change in the International prostate score system

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (2):
- Egypt (2):
  - Cairo university hospitals, Cairo
  - Kasr Alainy University Hospitals, Cairo